CLINICAL TRIAL: NCT04482738
Title: The Acute Response of Glucocorticoids Upon Food Intake
Brief Title: Study of the Effects of Overfeeding on Glucocorticoids in Lean and Obese Subjects
Acronym: Gluco-Food
Status: Completed | Type: Observational
Sponsor: Eleonora Seelig (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Eleonora Seelig, Principal Investigator, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: 202000384
Record Dates: First submitted 2020-03-30; First posted 2020-07-22 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Overweight and Obesity
Keywords: obesity; overweight; cortisol; overfeeding; glucocorticoids
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lean subjects: 24 hours before the study visit, participants will be asked to refrain from alcohol and strenuous exercise. Patients will be asked to remain fasted 10 hours before the study visit takes place. On the day of the study visit, patients will be admitted to the hospital and, after intake of the study meal, blood samples will be taken.
  Interventions: Other: High-calorie meal
- Obese subjects: 24 hours before the study visit, participants will be asked to refrain from alcohol and strenuous exercise. Patients will be asked to remain fasted 10 hours before the study visit takes place. On the day of the study visit, patients will be admitted to the hospital and, after intake of the study meal, blood samples will be taken.
  Interventions: Other: High-calorie meal

INTERVENTIONS:
Other: High-calorie meal — Intake of a high-calorie meal (2500-3000 calories) within 15 minutes.

SUMMARY:
Investigators suggest that in lean subjects cortisol increases in response to overfeeding and that this increase is blunted in obese subjects. A group of 18 male healthy lean subjects and another group of 18 male healthy obese subjects will undergo a high-calorie meal test. Prior to the meal intake, an indirect calorimetry, bioelectrical impedance, heart rate variability, a fasting blood sample and a perceived stress questionnaire will be assessed. After intake of the study meal, blood tests will be performed in order to measure the secretion of cortisol, glucose and lipid metabolism and inflammatory markers. Indirect calorimetry will be assessed again 60 and 180 minutes after the meal intake.

DETAILED DESCRIPTION:
Obesity is one of the most serious health problems in the 21st century. High energy food and a sedentary lifestyle are driving the current obesity pandemic. These factors activate the hypothalamic-pituitary-adrenal (HPA) axis, the key regulatory pathway of energy homeostasis. Activation of the HPA-axis leads to secretion of glucocorticoids from the adrenal glands, which control energy homeostasis by mobilizing and redistributing energy substrates.

Animal models of obesity have shown that glucocorticoids play a key role in the development of the metabolic syndrome. However, studies in humans yielded conflicting results. These studies have a major limitation in common. They do not consider glucocorticoid rhythmicity but rather investigate a snapshot of glucocorticoid secretion. Rhythmicity, however, is crucial because already minor glucocorticoid phase disturbances cause disease and could contribute to obesity.

Interestingly, excessive food intake may increase cortisol levels in healthy subjects . The consequence of this food-induced cortisol peak is not understood, but it may be key to restoring energy homeostasis after a meal. Whether the food-induced cortisol peak in obese subjects is disturbed is not known

With this study, investigators aim to better understand the role played by glucocorticoids in the origin of overweight and obesity. Researchers will investigate, in lean and obese subjects, whether the pulsatile release of cortisol increases after intake of a high-calorie meal. 36 subjects will take part in the study: a group of 18 male lean subjects and a second group of 18 male obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >18,5 and <25 kg/m2
* BMI >30 kg/m2

Exclusion Criteria:

* Any clinically significant concomitant diseases in lean subjects
* Any clinically significant concomitant diseases in obese subjects apart from features of the metabolic syndrome (dyslipidemia, arterial hypertension and insulin resistance)
* Lactose intolerance
* Severe food allergy
* Regular alcohol consumption (>30 g/d)
* Regular fitness training (>4 hours/week)
* Previous enrolment in a clinical trial within the last 3 months
* Inability or contradictions to undergo the investigated intervention
* Inability to follow the procedures of the study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample. The obese group will be both a community and a clinical sample.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Change in pulsatile secretion of cortisol in response to a high-calorie meal (nmol/l) | 195 minutes
  Blood test

SECONDARY OUTCOMES:
Thyroid hormones (nmol/l) | 195 minutes
  Blood test
Growth Hormone (mIU/l) | 195 minutes
  Blood test
Catecholamines (pg/ml) | 195 minutes
  Blood test
Adrenocorticotropic Hormone (ACTH) (pg/ml) | 195 minutes
  Blood test
Glucagon-like-peptide-1 (GLP-1) (pg/ml) | 195 minutes
  Blood test
Gastric inhibitory polypeptide (GIP) (pg/ml) | 195 minutes
  Blood test
Peptide YY (PYY) (pg/ml) | 195 minutes
  Blood test
Glucose (mmol/l) | 195 minutes
  Blood test
Insulin (mIU/l) | 195 minutes
  Blood test
C-Peptide (pmol/l) | 195 minutes
  Blood test
Total cholesterol (mmol/l) | 195 minutes
  Blood test
Low density lipoprotein (LDL)-cholesterol (mmol/l) | 195 minutes
  Blood test
High density lipoprotein (HDL)-cholesterol (mmol/l) | 195 minutes
  Blood test
Triglycerides (mmol/l) | 195 minutes
  Blood test
Growth differentiation factor 15 (GDF15) (ng/l) | 195 minutes
  Blood test
High-sensitive c-reactive Protein (hsCRP) (mg/l) | 195 minutes
  Blood test
Interleukin-6 (IL-6) (pg/ml) | 195 minutes
  Blood test
Interleukin-8 (IL-8) (pg/ml) | 195 minutes
  Blood test
Interleukin-1 receptor Antagonist (IL-1Ra) (pg/ml) | 195 minutes
  Blood test
Heart rate (bpm) | 5 minutes
  Heart rate variability analysis
Blood pressure: diastolic and systolic blood pressure (mmHg) | 1 minute
  Standard blood pressure monitor
Weight: kilogram body weight (kg) | 1 minute
  Standard scale
Energy expenditure: basal metabolic rate | 200 minutes
  Indirect calorimetry
Substrate utilisation: respiratory quotient | 200 minutes
  Indirect calorimetry
Fat and lean mass (kg) | 20 minutes
  Body impedance analysis
Total body water (l) | 20 minutes
  Body impedance analysis
Appetite: visual analogue scale rating | 3 hours
  Visual analogue scale
Stress: perceived stress Levels (0-56) | 5 minutes
  Perceived stress questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Seelig, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prospective Studies Collaboration; Whitlock G, Lewington S, Sherliker P, Clarke R, Emberson J, Halsey J, Qizilbash N, Collins R, Peto R. Body-mass index and cause-specific mortality in 900 000 adults: collaborative analyses of 57 prospective studies. Lancet. 2009 Mar 28;373(9669):1083-96. doi: 10.1016/S0140-6736(09)60318-4. Epub 2009 Mar 18. PMID 19299006
- [Background] van der Klaauw AA, Farooqi IS. The hunger genes: pathways to obesity. Cell. 2015 Mar 26;161(1):119-132. doi: 10.1016/j.cell.2015.03.008. PMID 25815990
- [Background] Vgontzas AN, Lin HM, Papaliaga M, Calhoun S, Vela-Bueno A, Chrousos GP, Bixler EO. Short sleep duration and obesity: the role of emotional stress and sleep disturbances. Int J Obes (Lond). 2008 May;32(5):801-9. doi: 10.1038/ijo.2008.4. Epub 2008 Feb 5. PMID 18253159
- [Background] de Guia RM, Rose AJ, Herzig S. Glucocorticoid hormones and energy homeostasis. Horm Mol Biol Clin Investig. 2014 Aug;19(2):117-28. doi: 10.1515/hmbci-2014-0021. PMID 25390020
- [Background] Russell G, Lightman S. The human stress response. Nat Rev Endocrinol. 2019 Sep;15(9):525-534. doi: 10.1038/s41574-019-0228-0. Epub 2019 Jun 27. PMID 31249398
- [Background] Ferrau F, Korbonits M. Metabolic Syndrome in Cushing's Syndrome Patients. Front Horm Res. 2018;49:85-103. doi: 10.1159/000486002. Epub 2018 Apr 5. PMID 29894989
- [Background] Livingstone DE, Grassick SL, Currie GL, Walker BR, Andrew R. Dysregulation of glucocorticoid metabolism in murine obesity: comparable effects of leptin resistance and deficiency. J Endocrinol. 2009 May;201(2):211-8. doi: 10.1677/JOE-09-0003. Epub 2009 Feb 17. PMID 19223399
- [Background] Livingstone DE, Jones GC, Smith K, Jamieson PM, Andrew R, Kenyon CJ, Walker BR. Understanding the role of glucocorticoids in obesity: tissue-specific alterations of corticosterone metabolism in obese Zucker rats. Endocrinology. 2000 Feb;141(2):560-3. doi: 10.1210/endo.141.2.7297. PMID 10650936
- [Background] Liu Y, Nakagawa Y, Wang Y, Li R, Li X, Ohzeki T, Friedman TC. Leptin activation of corticosterone production in hepatocytes may contribute to the reversal of obesity and hyperglycemia in leptin-deficient ob/ob mice. Diabetes. 2003 Jun;52(6):1409-16. doi: 10.2337/diabetes.52.6.1409. PMID 12765951
- [Background] Chalew S, Nagel H, Shore S. The hypothalamic-pituitary-adrenal axis in obesity. Obes Res. 1995 Jul;3(4):371-82. doi: 10.1002/j.1550-8528.1995.tb00163.x. PMID 8521154
- [Background] Marin P, Darin N, Amemiya T, Andersson B, Jern S, Bjorntorp P. Cortisol secretion in relation to body fat distribution in obese premenopausal women. Metabolism. 1992 Aug;41(8):882-6. doi: 10.1016/0026-0495(92)90171-6. PMID 1640867
- [Background] Duclos M, Corcuff JB, Etcheverry N, Rashedi M, Tabarin A, Roger P. Abdominal obesity increases overnight cortisol excretion. J Endocrinol Invest. 1999 Jun;22(6):465-71. doi: 10.1007/BF03343591. PMID 10435857
- [Background] Pasquali R, Cantobelli S, Casimirri F, Capelli M, Bortoluzzi L, Flamia R, Labate AM, Barbara L. The hypothalamic-pituitary-adrenal axis in obese women with different patterns of body fat distribution. J Clin Endocrinol Metab. 1993 Aug;77(2):341-6. doi: 10.1210/jcem.77.2.8393881.
- [Background] Chalew SA, Lozano RA, Armour KM, Zadik Z, Kowarski AA. Reduction of plasma cortisol levels in childhood obesity. J Pediatr. 1991 Nov;119(5):778-80. doi: 10.1016/s0022-3476(05)80302-6. No abstract available. PMID 1941386
- [Background] Chalew SA, Nagel H, Burt D, Edwards CR. The integrated concentration of cortisone is reduced in obese children. J Pediatr Endocrinol Metab. 1997 May-Jun;10(3):287-90. doi: 10.1515/JPEM.1997.10.3.287. PMID 9388820
- [Background] Jessop DS, Dallman MF, Fleming D, Lightman SL. Resistance to glucocorticoid feedback in obesity. J Clin Endocrinol Metab. 2001 Sep;86(9):4109-14. doi: 10.1210/jcem.86.9.7826. PMID 11549634
- [Background] Strain GW, Zumoff B, Strain JJ, Levin J, Fukushima DK. Cortisol production in obesity. Metabolism. 1980 Oct;29(10):980-5. doi: 10.1016/0026-0495(80)90043-8. PMID 6999293
- [Background] Pasquali R, Anconetani B, Chattat R, Biscotti M, Spinucci G, Casimirri F, Vicennati V, Carcello A, Labate AM. Hypothalamic-pituitary-adrenal axis activity and its relationship to the autonomic nervous system in women with visceral and subcutaneous obesity: effects of the corticotropin-releasing factor/arginine-vasopressin test and of stress. Metabolism. 1996 Mar;45(3):351-6. doi: 10.1016/s0026-0495(96)90290-5. PMID 8606643
- [Background] Rosmond R, Dallman MF, Bjorntorp P. Stress-related cortisol secretion in men: relationships with abdominal obesity and endocrine, metabolic and hemodynamic abnormalities. J Clin Endocrinol Metab. 1998 Jun;83(6):1853-9. doi: 10.1210/jcem.83.6.4843. PMID 9626108
- [Background] Longui CA, Giusti MM, Calliari LE, Katiki T, Kochi C, Monte O. Partial glucocorticoid resistance in obese children detected by very low dose dexamethasone suppression test. J Pediatr Endocrinol Metab. 2003 Dec;16(9):1277-82. doi: 10.1515/jpem.2003.16.9.1277. PMID 14714751
- [Background] Ljung T, Andersson B, Bengtsson BA, Bjorntorp P, Marin P. Inhibition of cortisol secretion by dexamethasone in relation to body fat distribution: a dose-response study. Obes Res. 1996 May;4(3):277-82. doi: 10.1002/j.1550-8528.1996.tb00546.x. PMID 8732962
- [Background] Woods C, Tomlinson JW. The Dehydrogenase Hypothesis. Adv Exp Med Biol. 2015;872:353-80. doi: 10.1007/978-1-4939-2895-8_16. PMID 26216003
- [Background] van Rossum EF. Obesity and cortisol: New perspectives on an old theme. Obesity (Silver Spring). 2017 Mar;25(3):500-501. doi: 10.1002/oby.21774. No abstract available. PMID 28229549
- [Background] Al-Damluji S, Iveson T, Thomas JM, Pendlebury DJ, Rees LH, Besser GM. Food-induced cortisol secretion is mediated by central alpha-1 adrenoceptor modulation of pituitary ACTH secretion. Clin Endocrinol (Oxf). 1987 May;26(5):629-36. doi: 10.1111/j.1365-2265.1987.tb00819.x. PMID 2822298
- [Background] Benedict C, Hallschmid M, Scheibner J, Niemeyer D, Schultes B, Merl V, Fehm HL, Born J, Kern W. Gut protein uptake and mechanisms of meal-induced cortisol release. J Clin Endocrinol Metab. 2005 Mar;90(3):1692-6. doi: 10.1210/jc.2004-1792. Epub 2004 Dec 7. PMID 15585568
- [Background] Follenius M, Brandenberger G, Hietter B. Diurnal cortisol peaks and their relationships to meals. J Clin Endocrinol Metab. 1982 Oct;55(4):757-61. doi: 10.1210/jcem-55-4-757. PMID 7202017
- [Background] Ibrahim M, Bonfiglio S, Schlogl M, Vinales KL, Piaggi P, Venti C, Walter M, Krakoff J, Thearle MS. Energy Expenditure and Hormone Responses in Humans After Overeating High-Fructose Corn Syrup Versus Whole-Wheat Foods. Obesity (Silver Spring). 2018 Jan;26(1):141-149. doi: 10.1002/oby.22068. Epub 2017 Nov 28. PMID 29193741
- [Background] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169